CLINICAL TRIAL: NCT04586179
Title: A Physiological and Clinical Comparison Between Cardiovascular Exercise Modes Following Sport Related Concussion
Brief Title: A Comparison Between Cardiovascular Exercise Modes Following Sport Related Concussion
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to enroll target number of participants.
Sponsor: University of Pittsburgh (Other)
Collaborators: University of Pittsburgh Medical Center (Other)
Responsible Party: Principal Investigator, Anthony P. Kontos, Ph.D., Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: STUDY20010091
Record Dates: First submitted 2020-09-29; First posted 2020-10-14 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2022-05

CONDITIONS: Concussion, Mild; Sport Injury
Keywords: sport-related concussion; concussion therapy; aerobic exercise; exercise testing
MeSH Terms: conditions — Brain Concussion | interventions — Exercise

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Care provider will not be aware of group assignment; participant will be aware of intervention assessment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic (treadmill) Exercise (Active Comparator): Participants will wear a heart rate monitor and complete the Buffalo Concussion Treadmill Test
  Interventions: Other: Aerobic (treadmill) Exercise
- Dynamic Exercise (Experimental): Participants will wear a heart rate monitor and complete a dynamic exertion assessment that incorporates directional changes that incrementally increases in exercise intensity
  Interventions: Other: Dynamic (Agility) Exercise

INTERVENTIONS:
Other: Aerobic (treadmill) Exercise — Individuals begin walking at 5.8 km/hr. (3.6 mph) at a 0.0% incline (5.1 km/hr. [3.2 mph] if below 5' 10" tall), the treadmill incline is increased 1 degree each minute for the first 15 minutes, then speed increased 0.64 km/hr. (0.4 mph) each minute thereafter.
  Exercise will be terminated if participant a) attains 90 percent of predicted heart rate reserve (HRR=.90*[{208-(.7*age)}-resting HR]), or b) reports a symptom worsening of 3 or points (0-10 scale) for headache, dizziness, or nausea, d) a rapid progression of complaints with continued exercise, or e) a rating of perceived exertion (RPE) greater than 18.5.
  Arms: Aerobic (treadmill) Exercise
Other: Dynamic (Agility) Exercise — Participants will begin in a center circle with equidistant cones 2.5 meters away. After the administrator presents a card, the participant touches a corresponding cone and returns to the starting position. Cards will be presented in increasing frequency in synchrony with a metronome application until exercise termination criteria are identified.
  Exercise will be terminated if participant a) attains 90 percent of predicted heart rate reserve (HRR=.90*[{208-(.7*age)}-resting HR]), or b) reports a symptom worsening of 3 or points (0-10 scale) for headache, dizziness, or nausea, d) a rapid progression of complaints with continued exercise, or e) a rating of perceived exertion greater than 18.5.
  Arms: Dynamic Exercise

SUMMARY:
Primary Aim: Compare physiological (e.g., heart rate) and clinical responses (e.g., symptom provocation) of adolescent and adult athletes (14-35 years of age) completing either a structured treadmill running or a dynamic aerobic exertion protocol during the subacute phase of sport-related concussion recovery (3-30 days after injury).

Secondary Aim: Examine potential effects of clinically-relevant factors that influence symptom responses to controlled aerobic exertion, such as age, physical activity patterns, motion sensitivities, psychological responses to injury, and sleep quality, among subjects completing controlled aerobic and dynamic exertion following sport-related concussion

DETAILED DESCRIPTION:
Exercise testing is an emerging component of the clinical evaluation for sport-related concussion. Despite the growing empirical evidence to suggest that early activity following an initial rest period after injury is beneficial to recovery, the effects of modifiable exercise prescription factors (e.g., exercise mode, duration, and intensity) is unknown. Given that dynamic exertion, which incorporates synchronized head-body movements, may contribute greater information processing demands for the functional pathways responsible for balance and equilibrium than treadmill running, may be more likely to provoke symptoms during exertion. Thus, physically active (>150 min/week of moderate-intensity physical activity) participants prior to a diagnosed sport-related concussion will be randomly assigned to complete either an aerobic or dynamic exercise task at 1 study visit following injury.

ELIGIBILITY:
Inclusion Criteria:

* Ages 14-35
* Prior to injury, participant fulfilled ACSM's guidelines for regular aerobic activity (30 minutes of moderate-intensity exercise 5 days per week or 20 minutes of vigorous exercise 3 days per week) prior to injury.
* Diagnosed with a sport related concussion within 14 days of injury in the window of 3-30 days prior to completing the first study visit, and also being a single episode.
* Participants referred to exertion therapy after a trained clinician from University of Pittsburgh Medical Center (UPMC) Sports Medicine Concussion Program has interpreted neurocognitive, vestibular, and clinical interview outcomes

Exclusion Criteria:

* History of brain surgery or traumatic brain injury(based on Glasgow Coma Scale of <13)
* History of neurological disorder (seizure disorder, epilepsy, brain tumors or malformations)
* Current history of pre-existing vestibular disorder [benign paroxysmal positional vertigo (BPPV), labyrinthitis or vestibular neuritis]
* Previous diagnosis of ocular motor condition (Ocular motor apraxia)Currently taking anticoagulant, beta-blockers, and anticonvulsant prescription medication
* Diagnosed with a cardiac, peripheral, or cerebrovascular disease (type 1 or 2 diabetes, or renal disease.
* Experienced chest pain or shortness of breath while at rest or with mild exertion.
* Lose balance because of dizziness or have lost consciousness (aside from concussion) from exertion
* Diagnosed with or taking medication for a chronic medical condition
* Currently have a mental or physical impairment exacerbated by physical activity, leading to the inability to complete 30 minutes of moderate to vigorous exercise
* Been told by a doctor to only conduct physical activity under medical supervision.

Ages: 14 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2020-09-27 (Actual); Primary Completion 2021-06-03 (Actual); Study Completion 2021-06-03 (Actual)

PRIMARY OUTCOMES:
Changes in Concussion Symptoms From Pre to Post Exercise | At 1 study visit within 30 days following concussion, and within 15 minutes of initiating exercise until approximately 15 minutes after exercise cessation
  Concussion symptoms will be measured with the Post-concussion Symptom Scale (PCSS), a patient-report survey of 22 concussion-associated symptoms on a 0-6 Likert scale (0 'none' to 6 'severe'). Number of reported symptoms (range: 0- 22) and total symptom severity (range: 0-132) whereby greater scores indicate worse symptom burden will be examined. The survey takes approximately 5 minutes to complete
Heart Rate | At 1 study visit within 30 days following concussion, and within 15 minutes of initiating exercise until approximately 15 minutes after exercise cessation
  Actual and percent of age-estimated heart rate, measured in beats per minute , will be recorded prior to (approximately 5 min), during, and following (approximately 5 min) exercise via a noninvasive heart rate monitor. Heart rate at rest, exercise cessation, and their difference (maximum heart rate - resting heart rate) will be recorded.
Systolic and Diastolic Blood Pressure | At 1 study visit within 30 days following concussion, and within 15 minutes of initiating exercise until approximately 15 minutes after exercise cessation
  Systolic and diastolic blood pressure, measured in mmHg with a non-invasive blood pressure cuff, will be recorded prior to and following exercise intervention.
Exercise duration | Completed during the 1 study visit within 30 days following concussion
  Exercise duration, the time interval between exercise initiation and cessation, will be recorded in seconds (range: 0-900)
Clinical recovery | Through study completion, approximately between 3 and 30 days following concussion
  Duration of clinical recovery, measured in days, is the interval between injury onset until medical clearance to resume unrestricted sport participation.

SECONDARY OUTCOMES:
Changes in vestibular ocular motor screening (VOMS) symptoms from pre-exercise to post-exercise | At 1 study visit within 30 days following concussion, and within 15 minutes of initiating exercise until approximately 15 minutes after exercise cessation
  The vestibular/ocular motor screening (VOMS) tool is a brief (approximately 5 minutes) patient-reported assessment to screen for vestibular and ocular motor impairments after concussion. Participants report on a 0-10 Likert scale (0 'none' to 10 'severe') prior to and following each of the 7 VOMS sub-tests: smooth pursuits, horizontal saccades, vertical saccades, near-point of convergence, horizontal vestibular-ocular reflex, vertical vestibular-ocular reflex, visual motion sensitivity; and near point of convergence (NPC) distance. Symptoms will be totaled across all symptoms and sub-tests (maximum=240) whereby greater scores indicate worse symptom burden.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony P Kontos, PhD, Study Director — UPMC Sports Medicine Concussion Program
Locations (1):
- Neuromuscular Research Laboratory-Warrior Human Performance Research Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Sharing Statement: Deidentified Individual participant data that underlie the current protocol will be available. Study protocol, statistical analysis plan, informed consent form, and individual participant data will be available (including data dictionary) beginning 12 months following completion of study and ending 36 months afterward. Investigators who provide a methodologically sound proposal to achieve individual participant data for meta-analyses should be directed to: https://www.nmrl.pitt.edu/ OR https://www.orthonet.pitt.edu/research/research-centers-and-labs/concussion-research-laboratory
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 months following completion of study and ending 36 months afterward
Access Criteria: Investigators who provide a methodologically sound proposal to achieve individual participant data for meta-analyses
URL: http://www.orthonet.pitt.edu/research/research-centers-and-labs/concussion-research-laboratory

REFERENCES:
- [Background] Orr R, Bogg T, Fyffe A, Lam LT, Browne GJ. Graded Exercise Testing Predicts Recovery Trajectory of Concussion in Children and Adolescents. Clin J Sport Med. 2021 Jan;31(1):23-30. doi: 10.1097/JSM.0000000000000683. PMID 30439726
- [Background] Lal A, Kolakowsky-Hayner SA, Ghajar J, Balamane M. The Effect of Physical Exercise After a Concussion: A Systematic Review and Meta-analysis. Am J Sports Med. 2018 Mar;46(3):743-752. doi: 10.1177/0363546517706137. Epub 2017 Jun 1. PMID 28570092
- [Background] Lumba-Brown A, Teramoto M, Bloom OJ, Brody D, Chesnutt J, Clugston JR, Collins M, Gioia G, Kontos A, Lal A, Sills A, Ghajar J. Concussion Guidelines Step 2: Evidence for Subtype Classification. Neurosurgery. 2020 Jan 1;86(1):2-13. doi: 10.1093/neuros/nyz332. PMID 31432081